CLINICAL TRIAL: NCT01834092
Title: Measurement of the Endothelial Function in Patients With a Abdominal Aortic Aneurism.
Brief Title: Study of the Glycocalyx in Abdominal Aortic Aneurysm
Acronym: Endo_eAAA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Thomas Bech Jorgensen, MD, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-4-2012-085
Record Dates: First submitted 2013-04-13; First posted 2013-04-17 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Abdominal Aortic Aneurism; Surgery; Ischemic Reperfusion Injury
Keywords: Abdominal Aortic Aneurism; Endothelia; Glycocalyx; Reperfusion; Plasma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fresh frozen plasma (Active Comparator): 2 portions of FFP will be transfused prior to reperfusion
  Interventions: Other: Plasma
- Fresh non-frozen plasma (Experimental): 2 portions of non-frozen plasma will be transfused prior to reperfusion
  Interventions: Other: Plasma

INTERVENTIONS:
Other: Plasma — 2 Units of plasma transfused equvilant to 2 times 275ml
  Other Names: Fresh frozen plasma versus fresh non-frozen plasma

SUMMARY:
The investigators want to measure the degradation of the endothelial glycocalyx before and after clamping the aorta, in patients operated for a abdominal aortic aneurism.

DETAILED DESCRIPTION:
50 patients is scheduled for enrollment. Blood samples will be up taken before surgery, 10 min after reperfusion, at the end of surgery and the following morning. In addition the investigators are placing a renal venous catheter where blood samples will be up taken as mentioned above for the analysis of endothelial markers together with markers for kidney damage.

The first 10 patient will act as part of a pilot study, where only measurement of the endothelial and renal failure markers will be performed.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years

Exclusion Criteria:

* prior engagement in scientific study within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Endothelial dysfunction | 24 hours
  Measurement of endothelial markers peri- and postoperative: thrombomodulin, E-selectin and syndecan-1

SECONDARY OUTCOMES:
Fluid balance | 24 hours
  Perioperative and postoperative first 24 hours

OTHER OUTCOMES:
Postoperative organ failure | 30 days
  Development of kidney- and respiratory failure and sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Per I Johansson, MD, Study Chair — Section for Transfusion Medicine, Capital Region Blood Bank, Rigshospitalet, Copenhagen, Denmark.
Locations (1):
- Rigshospitalet, Copenhagen, Østerbro, Denmark